CLINICAL TRIAL: NCT04103970
Title: The Effect of Graded Activity and Pain Education (GAPE) for Patients Early After Lumbar Spinal Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Frederiksberg University Hospital (Other); Defactum, Central Denmark Region (Other Government)
Responsible Party: Principal Investigator, Heidi Tegner, Principal Investigator, PT, MScH, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-19024440
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2023-11

CONDITIONS: Low Back Pain
Keywords: Low back pain; Back surgery; Lumbar spinal fusion; Postoperative rehabilitation; Graded activity; Pain education; Disability; Pain; Fear of movement; Self-efficacy for exercise; Health related quality of life; Sedentary behavior
MeSH Terms: conditions — Low Back Pain; Pain; Kinesiophobia; Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Usual care:
  Before surgery all patients are invited to participate in a pre-surgery seminar, where they receive information and advice about the time before, during and after the LSF. The seminar will be guided by nurses, surgeons, anesthesiologist, occupational therapists and physiotherapist.
  After the surgery the patient will be hospitalized on an average of 3-4 days. During hospitalization a physiotherapist consults the patients on a daily basis to provide information, guidance on mobilization and instructions in gradually progressing movement. The patients will have no restrictions on movement after surgery and should gradually return to normal activity level.
  Three months post-operatively all patients will receive physical rehabilitation delivered by physiotherapists in a community care center.
- Intervention group: Graded Activity and Pain Education (GAPE) (Experimental): Patients in the intervention-group will receive usual care and 9 sessions of GAPE, 4 sessions at the hospital, 2 sessions in the patient's home and 3 sessions by telephone.
  Pain education in GAPE is viewed as an approach which target cognitive attitudes and beliefs about pain. The pain education will target 3 overall questions: 1. What is pain and is my pain normal? 2. What can affect my pain? 3. What can I do to relieve my pain? The education will be individually adjusted to each patient, so the patient's context and concerns regarding pain and movement are included.
  The aim of Graded activity is to improve the patient's functional ability by positive reinforcement of health behaviors and activity levels. Graded activity will be based on which short-term activity-goals the patient evaluates as the most important for the treatment outcome. In close collaboration with the patient the physiotherapist will set quotas for the selected exercises/activities.
  Interventions: Behavioral: Graded Activity and Pain Education (GAPE)

INTERVENTIONS:
Behavioral: Graded Activity and Pain Education (GAPE) — GAPE is based on a cognitive behavioral perspective that human behavior is affected by behavioral, cognitive and affective factors, this include the patient's perception of and response to pain. The perspective is a psycho-social perspective which amplify and interact with the individual patient's pathology.
  The overall theoretical perspective in GAPE is that fear of movement and/or lack of self-efficacy for exercise can potentially lead to disuse and sedentary behavior, a perspective modified from the fear-avoidance model. In this modified version the patients´ and the physiotherapists´ former experiences, knowledge, and beliefs are factors influencing on the patients´ experience of pain and thereby their self-efficacy for exercise and fear of movement.
  Arms: Intervention group: Graded Activity and Pain Education (GAPE)

SUMMARY:
Background An increasing number of patients with chronic low back pain (CLBP) undergo lumbar spinal fusion (LSF). Unfortunately, a substantial part of the patients still has persistent pain, functional disability and poor quality of life after surgery. Research in the field of rehabilitation after LSF call for high quality research to focus on active approaches which incorporate an early bio-psycho-social focus. A focus which include the patient's context, experiences and thoughts even more in the clinical decision making.

The primary objective of this trial is to examine the effect of an early active rehabilitation-intervention consisting of Graded Activity and Pain Education (GAPE) on sedentary behavior in a population of patients undergoing LSF. The secondary objectives are to examine the effect of GAPE on disability, pain, fear of move-ment, self-efficacy for exercise and health related quality of life.

Methods:

The study is a randomized controlled trial planned to include 144 patients after LSF caused by degeneration of the lumbar spine (including spondylolisthesis). The patients will be randomly assigned to receive either usual care or usual care plus GAPE. GAPE consists of 9 individual sessions, with an overall purpose to influence the patient beliefs and thoughts about movement and pain towards increased self-efficacy for exercise and decreased fear of movement. A physiotherapist will in close collaboration with the patient plan GAPE based on an in-depth pain-anamnesis, individually set functional goals and observations of the patients in their homes. The primary outcome will be "reduction in sedentary behavior" measured by an accelerometer. Sec-ondary outcome will include disability, pain, fear of movement, self-efficacy for exercise and quality of life. Data will be collected at baseline (pre-surgery), and at 3, 6- and 12-months post-surgery.

DETAILED DESCRIPTION:
Introduction:

Over half a Billion people worldwide report low back pain (LBP), and it is the leading cause of disability at all levels of income and age groups. For the majority of people with LBP the condition has a natural course and the pain will diminish over time, but for a small percentage the conditions turns into a chronic state with significant levels of life disruption, healthcare costs and economic losses and even premature death. Lumbar spinal fusion (LSF) is a widely adopted surgical procedure for the treatment of persistent LBP, with the aim of relieving pain and increasing functional ability. Over recent decades a substantially increasing number of patients with chronic low back pain (CLBP) undergo LSF in the western world.

Unfortunately, a substantial part of the patients undergoing spine surgery still have persistent pain, functional disability and poor quality of life 4 and 8-10 years after surgery. A report from the Swedish Spine register shows that pain level remains the same 1-5 years after LSF for 25 % of the patients, and consumption of medication remains unchanged in almost 50 % of the patients.

Rationale:

The majority of patients (70 %) planned for spine surgery have fear of movement, and it is well supported in the literature that fear of movement, avoidance coping, negative affect and depression postoperative are associated with persistent pain and function after spine surgery up to 3 years postoperative. Individual differences of pain related coping strategies after LSF also seems to have an influence on the patient's sedentary behavior postoperative.

Research in the field of rehabilitation after LSF have thereby resulted in a growing consensus that a bio-psycho-social approach to rehabilitation is needed. An approach which should start quite early after surgery, and which should focus on the patient's diverse way of living with a disease and the interrelationship between both the biological, psychological and social factors.

A systematic review found that "complex interventions" comprising of exercise and cognitive behavioral therapy offers short and long term functional benefits to patients following LSF. Another RCT confirmed that an early intervention using a cognitive behavioral approach performed by a physiotherapist decreased fear of movement, increased self-efficacy and improved patient-reported and performance-based outcomes in patients after lumbar spine surgery six months after surgery. Research in the field of rehabilitation after LSF call for high quality research to confirm the importance of including an early active approach with a cognitive and behavioral perspective, and advocate for interventions to incorporate the patients context, experiences and thoughts even more in the clinical decision making.

Intervention:

Graded activity is an exercise paradigm which takes a behavioral approach using the principles of operant conditioning. The principles of operant conditioning are to modify negative pain behaviors and disrupt the fear avoidance cycle and thereby increase the patient's physical activity or functioning. Relevant information about pain, healing and the effects of disuse can likely influence what a patient anticipate about movement despite pain. Several studies have investigated the effect of pain education to patients with CLBP and found it efficient. A combination of pain education and exercise for patients with CLBP are furthermore showing promising results. Therefore, a combination of Graded Activity and Pain Education (GAPE) seems to be a suitable approach for early post-operative rehabilitation for patients with LSF, as behavioral, cognitive and physical factors will be addressed in one intervention.

Objective and hypothesis The primary objective of this randomized controlled trial is to examine the effect of an early active intervention consisting of Graded Activity and Pain Education (GAPE) on sedentary behavior in a population of patients undergoing LSF. The secondary objectives are to examine the effect of GAPE on disability, pain, fear of movement, self-efficacy for exercise and health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

Patients from the Capital Region of Denmark undergoing LSF at Centre for Rheumatology and Spine Diseases, Rigshospitalet, Glostrup from 23st of September 2019 to 30st marts 2021 and fulfilling the following criteria:

1. Low back pain > six months
2. >18 years
3. Undergoing an instrumented spinal posterior fusion of 1-2 spinal segments for degeneration of the lumbar spine, with or without an intervertebral cage placed from the anterior approach, posterior approach or from a lateral access.

   Degenerative conditions include disc herniation, spinal stenosis, spondylosis with or with-out myelopathy and spondylolisthesis.
4. Read and understand Danish
5. Lives no more than 1 ½ hour of transportation from Rigshospitalet, Glostrup

Exclusion Criteria:

1. Has previously been through an LSF
2. One or more of following conditions (infection, neoplasm, metastasis, metabolic bone dis-ease, fractures, post-traumatic vertebral compression/deformity or other known autoimmune arthropathies)
3. Are cognitively or otherwise unable to give informed consent and adhere to the study program
4. Other special conditions where a patient is judged not able to participate in the intervention by the surgeon or researcher (HT) (weakness caused by very high age, extreme poorly functional level, other serious comorbidities)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sedentary behavior (sitting or reclining/lying posture) | 3 months post-surgery
  Sedentary behavior will in this study be defined as: "Any waking behavior characterized by a sitting or reclining/lying posture". Sedentary behavior will be assessed objectively as the number of minutes per day the patient is sedentary (lying down and sitting) measured by SENS motion activity measurement system. SENS is a small accelerometer placed within a small plaster to be worn on the patient's thigh. The SENS motion system is considered a reliable and valid device for measuring sedentary behavior. The patients will wear the accelerometer for 7 consecutive days during the week before surgery, and in 7 days at three- and 12-months post-surgery.

SECONDARY OUTCOMES:
Change from baseline in sedentary behavior (sitting or reclining/lying posture) | 12 months
  Sedentary behavior will in this study be defined as: "Any waking behavior characterized by a sitting or reclining/lying posture". Sedentary behavior will be assessed objectively as the number of minutes per day the patient is sedentary (lying down and sitting) measured by SENS motion activity measurement system. SENS is a small accelerometer placed within a small plaster to be worn on the patient's thigh. The SENS motion system is considered a reliable and valid device for measuring sedentary behavior. The patients will wear the accelerometer for 7 consecutive days during the week before surgery, and in 7 days at three- and 12-months post-surgery.
Ostwestry Disability Index: Disability | Baseline, 3, 6 and 12 months post-surgery
  Disability will be measured using the Oswestry Disability Index (ODI). ODI is a validated measure of condition-specific disability originally developed for patients with LBP. The Danish version of ODI has been validated and shown acceptable responsiveness, reliability, and validity. The ODI consists of ten items regarding pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and traveling. For each item the patient chooses one of six answers, with 0 representing no difficulty in the activity and 5 representing maximal difficulty.
Visual Analogue Scale (VAS pain): Pain | Baseline, 3, 6 and 12 months post-surgery
  Pain in the back and legs is assessed using a visual analogue scale (VAS). The endings of the line have verbal descriptions: 0 (''no pain'') - 100 ("the worst pain imaginable"). An example of a VAS scale is drawn and the text to the scale is as following: "Mark your pain level for the past week by a mark on each line below as in the example. The lines are a scale that on the far left corresponds to painless and on the far right corresponds to the worst possible pain. With a mark on the line you register how your pain has been within the past week".
Tampa scale of Kinesiophobia: Fear of movement | Baseline, 3, 6 and 12 months post-surgery
  Fear of movement will be assessed using the Tampa Scale of Kinesiophobia (TSK). The TSK has shown satisfactory psychometric properties and validity in a wide variety of spinal and musculoskeletal diseases, including neck pain, LBP, and fibromyalgia. TSK is also a responsive measure in subjects after lumbar fusion undergoing multidisciplinary cognitive behavioral rehabilitation. The original version of TSK consisted of 17 items intended to assess fear of movement and fear of (re)injury. In this study a short version of 11 items will be used, as this has also been found valid, reliable and responsive. Respondents are asked to indicate to what extent the items are a true description of the assumed association between movement and (re)injury on a 4-point Likert scale, ranging from strongly disagree to strongly agree. Several studies have found support for the construct and predictive validity and reliability.
EuroQol 5: Health-related quality of life | Baseline, 3, 6 and 12 months post-surgery
  Quality of life will be assessed using the EuroQol 5 Dimensions 3 levels (EQ-5D-3L). The EQ-5D is a generic questionnaire developed by an international research group including researchers from Denmark. EQ-5D-3L consist of 5 dimensions in health-related quality of life: Mobility, Self-care, usual activities, Pain/discomfort, and anxiety/depression. Each dimension is divided into three levels: no problems, some problems or extreme problems. EQ-5D-3L also include a 20-cm vertical scale, were the respondent are asked to describe his/her own health with endpoints of 'best imaginable health state' set at 100 and 'worst imaginable health state' set at 0. The EQ-5D has been validated in Danish, including the development of preference values and Danish population norms.
Self-efficacy for exercise scale: Self-efficacy for exercise | Baseline, 3, 6 and 12 months post-surgery
  Self-efficacy for exercise will be assessed using the questionnaire Self-efficacy for Exercise Scale (SEES). The SEES consist of nine items that measure how confident the patient is in exercising. The total range is from 0 to 90 points were higher scores indicate a higher degree of self-efficacy for exercise. The SEES is translated to Swedish and show substantial test-retest reliability and satisfactory content and internal consistency with older adults. SEES included in this study will be a Danish (not validated) version of SEES.
Patient satisfaction with results of the surgery | Baseline, 3, 6 and 12 months post-surgery
  Patient satisfaction will be used to evaluate the patient's satisfaction regarding movement and pain after surgery.
  Regarding movement patients will be asked to judge their capacity to move their back after surgery on a visual analogue scale (VAS). In their considerations they are asked to include both movement of the back during activity of daily living and how safe they feel during movement of their back. The endings of the line have verbal descriptions: 0 (''very satisfied with my capacity to move my back post-surgery'') - 100 ("Not at all satisfied with my capacity to move my back post-surgery").
  Regarding pain patients will be asked to compare back/leg pain before operation until now. The patient can mark in 5 boxes from: "The pain is disappeared" to "The pain is worsened" The patient will also be asked to judge the overall result of the operation from "Satisfied" to "Not satisfied".

CONTACTS AND LOCATIONS:
Overall Officials: Marius Henriksen, Study Chair — Faculty of Health Sciences, Copenhagen University
Locations (1):
- Department of Occupational and Physiotherapy, Rigshospitalet Glostrup, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tegner H, Rolving N, Henriksen M, Bech-Azeddine R, Lundberg M, Esbensen BA. The Effect of Graded Activity and Pain Education After Lumbar Spinal Fusion on Sedentary Behavior 3 and 12 Months Postsurgery: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2024 Aug;105(8):1480-1489. doi: 10.1016/j.apmr.2024.04.005. Epub 2024 Apr 27. PMID 38685291
- [Derived] Tegner H, Esbensen BA, Henriksen M, Bech-Azeddine R, Lundberg M, Nielsen L, Rolving N. The effect of graded activity and pain education (GAPE): an early post-surgical rehabilitation programme after lumbar spinal fusion-study protocol for a randomized controlled trial. Trials. 2020 Sep 15;21(1):791. doi: 10.1186/s13063-020-04719-y. PMID 32933571